CLINICAL TRIAL: NCT03379376
Title: EHealth Mindful Movement and Breathing to Improve Gynecologic Cancer Surgery Outcomes: Aim II
Brief Title: EHealth Mindful Movement and Breathing in Improving Outcomes in Participants Undergoing Gynecologic Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Wake Forest University Health Sciences (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: IRB00046462; NCI-2018-00584 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); CCCWFU 04517 (Other: Wake Forest University Health Sciences); P30CA012197 (NIH)
Record Dates: First submitted 2017-11-29; First posted 2017-12-20 (Actual); Results first posted 2019-12-23 (Actual); Last update posted 2019-12-30 (Actual); Status verified 2019-12

CONDITIONS: Female Reproductive System Neoplasm; Malignant Female Reproductive System Neoplasm; Malignant Uterine Neoplasm; Ovarian Carcinoma; Ovarian Neoplasm; Suspicious for Malignancy; Uterine Neoplasm
MeSH Terms: conditions — Genital Neoplasms, Female; Uterine Neoplasms; Ovarian Neoplasms | interventions — Palliative Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Supportive Care (eMMB) (Experimental): Participants receive a self-directed 20-minute eMMB video and are instructed to practice eMMB at least once before surgery and daily for 2 weeks after surgery. Participants may also request additional guidance from a yoga instructor via telephone and video conference before surgery and again 1 day after surgery or as soon as feasible.
  Interventions: Other: Questionnaire Administration; Procedure: Supportive Care

INTERVENTIONS:
Other: Questionnaire Administration — Receive questionnaire
Procedure: Supportive Care — Undergo eHealth mindful moving and breathing
  Other Names: Supportive Therapy; Symptom Management; Therapy, Supportive

SUMMARY:
This trial determines how well eHealth mindful movement and breathing works to improve outcomes in participants undergoing gynecologic surgery. Supportive therapy, such as eHealth mindful movement and breathing, uses techniques that include gentle movements, breathing, and relaxation techniques which may help participants cope with and improve their surgical experiences.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To field-test implementation strategies of the mindful movement and breathing (eMMB) intervention that has been adapted to the eHealth Format.

OUTLINE:

Participants receive a self-directed 20-minute eMMB video and are instructed to practice eMMB at least once before surgery and daily for 2 weeks after surgery. Participants may also request additional guidance from a yoga instructor via telephone and video conference before surgery and again 1 day after surgery or as soon as feasible.

After completion of study, participants are followed up at 4 weeks from surgery.

ELIGIBILITY:
Inclusion Criteria:

* Scheduled for an abdominal gynecological surgery (i.e. uterine, ovarian) to remove a mass that is suspected to be malignant
* Have an Eastern Cooperative Oncology Group (ECOG) performance status of ≤1
* Cognitively able to complete assessments as judged by the study team
* Able to understand, read and write English

Exclusion Criteria:

* Have schizophrenia or any other psychotic disorder
* Have a diagnosed sleep disorder including untreated obstructive sleep apnea, periodic limb movement disorder, or restless leg syndrome

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2018-04-05 (Actual); Primary Completion 2018-10-15 (Actual); Study Completion 2018-11-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Stephanie Sohl, Principal Investigator — Wake Forest University Health Sciences
Locations (1):
- Wake Forest University Health Sciences, Winston-Salem, North Carolina, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Supportive Care (eMMB)
Started | 10
Completed | 5
Not Completed | 5
Not completed — Lost to Follow-up | 2
Not completed — Did not wish to complete follow up | 1
Not completed — Overwhelmed, didn't want to continue | 1
Not completed — Death | 1

BASELINE CHARACTERISTICS:
Arm/Group | Supportive Care (eMMB)
Number analyzed (Participants) | 10
Age, Continuous [Mean (Standard Deviation); unit: Years] | 58.2 (14.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10
  Male | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 10
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 8
  More than one race | 1
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 10

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Confident in the Use of EHealth Format
Description: This is a feasibility study to iteratively refine the eMMB implementation strategies with 10-15 consecutive participants enrolled. Participants will be asked to complete a brief usability questionnaire about their confidence in their ability to complete the intervention. The number of participants will depend on when a consensus is reached on a manual for implementing interventions and will be determined by calculating 95% confidence intervals around all the secondary outcomes.
Time Frame: Up to 4 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Supportive Care (eMMB)
Number analyzed (Participants) | 10
Participants | 7

2. Secondary Outcome: Number of Participants Recruited and Completed All Assessments
Description: Participants who were recruited and agreed to participate in the Mindful Movement and Breathing (eMMB) sessions and those who completed all assessments will be computed.
Time Frame: Up to 4 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Supportive Care (eMMB)
Number analyzed (Participants) | 10
Participants | 5

3. Secondary Outcome: Number of Participants That Adhered to Study Interventions
Description: To be determined by comparing participants who were adherent to attending study visits and interventions by an adherence assessment (1) Completion of the videoconference session; (2) any additional contact with the interventionists; (3) use of the self-directed intervention:
Time Frame: Up to 4 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Supportive Care (eMMB)
Number analyzed (Participants) | 10
Participants | 7

4. Secondary Outcome: Number of Participants Reporting Adverse Events
Description: Adverse events will be reported upon occurrence monthly. Specifically, they will be labeled definitely unrelated, definitely related, probably related, or possibly related to the study intervention.
Time Frame: Up to 4 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Supportive Care (eMMB)
Number analyzed (Participants) | 10
Participants | 1

5. Secondary Outcome: Percentage of Participants Completing 4-week Visits
Description: To be assessed by calculating the percent of participants who complete the 4-week visit.
Time Frame: Up to 4 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Supportive Care (eMMB)
Number analyzed (Participants) | 10
Participants | 5

ADVERSE EVENTS:
Time Frame: Nonserious adverse events will be monitored on a quarterly basis and serious adverse events up to 4 weeks.
Arm/Group | Supportive Care (eMMB)
All-Cause Mortality (participants affected / at risk) | 1/10
Serious Adverse Events (participants affected / at risk) | 1/10
Other Adverse Events (participants affected / at risk) | 0/10
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Supportive Care (eMMB) (N=10)
Sepsis (Infections and infestations) | 1 (1) — Led to death

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-04-20): https://cdn.clinicaltrials.gov/large-docs/76/NCT03379376/Prot_SAP_000.pdf